CLINICAL TRIAL: NCT05255887
Title: The Effect of Informing Patients With Video on Intensive Care Experiences Before Heart Surgery
Brief Title: The Effect of Informing Patients With Video Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Figen Dıgın, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KırklareliUU
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cardiovasculary Surgery, Education, Critical Care
Keywords: Cardiovascular surgery, education, critical care
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informing patients group (Experimental): 24-48 hours before the surgery, the patients will be shown an informative video about the intensive care environment in a separate room through a one-on-one interview. In the study, the day of discharge from the intensive care unit will be counted as the first day, and on the second day, the 'Intensive Care Experience Scale' will be applied to the patients in the experimental group by face-to-face interview method.
  Interventions: Other: Informing Patients With Video
- Control Group (No Intervention): patients who were no intervation

INTERVENTIONS:
Other: Informing Patients With Video — 24-48 hours before the surgery, the patients will be shown an informative video about the intensive care environment in a separate room through a one-on-one interview. (The content of the training to be done with the video is stated in the appendix) In the study, no attempt will be made to the control group patients other than the routine practice of the institution before the surgery. In the study, the day of discharge from the intensive care unit will be counted as the first day, and on the second day, the 'Intensive Care Experience Scale' will be applied to the patients in both the experimental and control groups by face-to-face interview method.
  Arms: Informing patients group

SUMMARY:
Purpose of the research; The aim of this study is to determine the effect of informing patients with video before heart surgery on their intensive care experience."Patient Descriptive Information Form" and "Intensive Care Experience Scale (ICES)" will be used to collect data.In Kavuncu's study, the average score they got from ICES was found to be 57.07±5.6. It was calculated that 45 patients from each group should be included in the study in order to test the 0.6-unit effect size value, which was calculated by accepting a 5% difference from this score in the experimental group, with a 5% margin of error, 95% confidence level and 80% power value.In the study, after the patients admitted to the cardiovascular surgery service for cardiac surgery were informed about the purpose and importance of the study and the research, informed consent will be obtained verbally and in writing from the volunteer patients. In order to ensure randomization of the patients in the study, a randomization plan was prepared for 45 experiments and 45 controls using a probabilistic scheme-based computer program.

DETAILED DESCRIPTION:
Purpose of the research; The aim of this study is to determine the effect of informing patients with video before heart surgery on their intensive care experience."Patient Descriptive Information Form" and "Intensive Care Experience Scale (ICES)" will be used to collect data.In Kavuncu's study, the average score they got from ICES was found to be 57.07±5.6. It was calculated that 45 patients from each group should be included in the study in order to test the 0.6-unit effect size value, which was calculated by accepting a 5% difference from this score in the experimental group, with a 5% margin of error, 95% confidence level and 80% power value.In the study, after the patients admitted to the cardiovascular surgery service for cardiac surgery were informed about the purpose and importance of the study and the research, informed consent will be obtained verbally and in writing from the volunteer patients. In order to ensure randomization of the patients in the study, a randomization plan was prepared for 45 experiments and 45 controls using a probabilistic scheme-based computer program. 24-48 hours before the surgery, the patients will be shown an informative video about the intensive care environment in a separate room through a one-on-one interview. In the study, no attempt will be made to the control group patients other than the routine practice of the institution before the surgery. In the study, the day of discharge from the intensive care unit will be counted as the first day, and on the second day, the 'Intensive Care Experience Scale' will be applied to the patients in both the experimental and control groups by face-to-face interview method.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above, open to communication and cooperation,
* He will have planned heart surgery,
* He is sane,
* Not having a diagnosis of psychiatric disease or using psychiatric medication,
* Do not have sensory problems such as vision, hearing and speech,
* Literate,
* speaking Turkish,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Under the age of 18 and not open to communication and cooperation,
* Unplanned or emergency heart surgery,
* mentally ill
* Diagnosed with psychiatric illness and using psychiatric medication,
* Having sensory problems such as vision, hearing and speech
* Being illiterate
* Does not speak Turkish,
* Patients who did not volunteer to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female patients will be included in the study.
Enrollment: 90 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
The effect of preoperative video training on patients' intensive care experience | 1 year
  The Intensive Care Experience Scale will be used for determining the effect of preoperative video training on patients' intensive care experience. According to 19 items with scale, the individual may determine his or her experiences in intensive care unit. The Intensive Care Experiences Scale are scored between 19 and 95. The lowest score that can be obtained from the scale is 19, the highest score is 95. As the total score obtained from the scale increases, it is evaluated that the patient's experience is positive and his awareness is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kalkan A, Digin F. The effect of informing patients with video before cardiac surgery on intensive care experience: A randomized controlled trial. Pak J Med Sci. 2024 Jul;40(6):1067-1072. doi: 10.12669/pjms.40.6.8627. PMID 38952513